CLINICAL TRIAL: NCT01576107
Title: Motivational Intervention Enhancing Physical Activity In Oncology Patients (MOTIVACTION)
Brief Title: MOTIVACTION - Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCT-PA8
Record Dates: First submitted 2012-04-05; First posted 2012-04-12 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Cancer
Keywords: Different cancer entities
MeSH Terms: conditions — Neoplasms | interventions — Behavior Therapy

ARMS (2):
- Physical activity (Experimental): Exercise counseling (behavior change techniques)
  Interventions: Other: Exercise counseling (behavior change techniques)
- Stress-management (Experimental): Stress-management training
  Interventions: Other: Stress-management training

INTERVENTIONS:
Other: Exercise counseling (behavior change techniques) — 4-week exercise intervention for cancer patients of different entities and out-patient regimes.
  Arms: Physical activity
Other: Stress-management training — 4-week stress-management-training for cancer patients of different entities and out-patient regimes.
  Arms: Stress-management

SUMMARY:
Impact of a 4-week exercise intervention vs. a stress-management-training on physical activity (measured objectively and by questionnaire) of cancer patients of different entities and out-patient regimes.

ELIGIBILITY:
Inclusion Criteria:

* Physical activity < 150 minutes /week
* Patients are currently receiving outpatient treatment (acute or maintenance therapy) or finished this therapy not longer than six months ago

Exclusion Criteria:

* Serious Orthopedic limitations
* Serious neurological disorders
* Serious cardiovascular diseases
* Bone metastases
* wound healing / scarring not completed
* Rehabilitation during the next eight weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Physical activity (accelerometer, Actigraph) | 4 weeks
  measured for 7 days

SECONDARY OUTCOMES:
physical activity (Short QUestionnaire to ASsess Healthenhancing physical activity, SQUASH) | 4 weeks, 3 months
  Wendel-Vos, G.C.W. et al., 2003
Self-Efficacy for Managing Chronic Disease 6-Item Scale (SES6G) | 4 weeks, 3 months
  German version by Freud, T. (2011)
Quality of life (EORTC QLQ C30) | 4 weeks, 3 months
  Aaronson, N. K. et al. (1993)
variables of the Health Action Process Approach | 4 weeks, 3 months
  scales are developed according to the guidelines by the founder of the theory (Schwarzer, 2008)
Barriers and barrier management in physical exercise | 4 weeks, 3 months
  adapted from Krämer&Fuchs (2010), developed in pilot studies
Exercise experience | 4 weeks, 3 Months
  questionnaire adapted from Fuchs, R., 2009

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wiskemann, Dr., Principal Investigator — German Cancer Research Center
Locations (2):
- Germany (2):
  - National Center for Tumor Diseases (German Cancer Research Center), Heidelberg, Baden-Wurttemberg
  - National Center for Tumor Diseases, Heidelberg, Baden-Wurttemberg

REFERENCES:
- [Derived] Ungar N, Wiskemann J, Sieverding M. Physical Activity Enjoyment and Self-Efficacy As Predictors of Cancer Patients' Physical Activity Level. Front Psychol. 2016 Jun 21;7:898. doi: 10.3389/fpsyg.2016.00898. eCollection 2016. PMID 27445882